CLINICAL TRIAL: NCT06623331
Title: The Implementation of Computer-aided Detection in an Initial Endoscopy Training Improves the Quality Measures of Trainees' Future Colonoscopies
Brief Title: The Implementation of Computer-aided Detection in Training Improves the Quality of Future Colonoscopies
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Zofia Orzeszko, Principal Investigator, Jagiellonian University
Other Study IDs: 2024.000.367
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Quality Indicators, Health Care; Colonoscopy Diagnostic Techniques and Procedures; Artificial Intelligence (AI)
Keywords: Quality Indicators; Colonoscopy; Artificial Intelligence (AI); Computer-aided detection (CADe); Adenoma detection rate (ADR)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Colonoscopies performed by endoscopists trained in AI-enhanced environment. The quality indicators are measured after completing training without AI enhancement.
  Interventions: Other: AI-enhanced endoscopy training
- Group B: Colonoscopies performed by endoscopists trained conventionally. The quality indicators are measured after completing training without AI enhancement.
  Interventions: Other: Conventional endoscopy training

INTERVENTIONS:
Other: AI-enhanced endoscopy training — Endoscopists trained in AI-enhanced environment. Their quality indicators are measured after completing training, without additional AI enhancement.
  Groups: Group A
Other: Conventional endoscopy training — Endoscopists trained conventionally
  Groups: Group B

SUMMARY:
Computer-aided detection (CADe) based on artificial intelligence (AI) may improve colonoscopy quality. An increasing number of young endoscopists are trained in an AI environment. However its impact on trainees' future outcomes remains unclear. The study aimed to evaluate the quality indicators of endoscopists trained in an AI environment compared to those trained conventionally.

DETAILED DESCRIPTION:
Computer-aided detection (CADe) based on artificial intelligence (AI) may improve colonoscopy quality. An increasing number of young endoscopists are trained in an AI environment. However its impact on trainees' future outcomes remains unclear. The study aimed to evaluate the quality indicators of endoscopists trained in an AI environment compared to those trained conventionally. A study included 6,000 adult patients who underwent a colonoscopy for various reasons. The study retrospectively evaluated the first 1,000 procedures performed by six endoscopists after completing training relying entirely on endoscopists' detection skills without AI enhancement. Three of those young endoscopists were trained with CADe, and three without additional assistance. Quality indicators were assessed in both groups. The morphology of detected polyps was evaluated to determine the influence of AI-enhanced training on laterally spreading tumors (LST) detection rate.

ELIGIBILITY:
Inclusion Criteria:

* adult participants who underwent a colonoscopy for various reasons performed by specific endoscopists that were assessed in terms of quality indicators

Exclusion Criteria:

* a history of bowel resection
* confirmed inflammatory bowel disease
* suspicion of polyps or cancer in other imaging tests
* suspicion of familial adenomatous polyposis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 6,000 adult patients who underwent a colonoscopy for various reasons in a single high-volume endoscopy clinic in Krakow.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Serrated polyp detection rate (SDR) | During the colonoscopy examination
  The percentage of colonoscopies when the serrated polyp was found
withdrawal time | During the colonoscopy examination
  The time from the cecal intubation to the end of the examination
Cecal intubation rate (CIR) | During the colonoscopy examination
  The percentage of colonoscopies with successful cecal intubations
Adenoma Detection Rate (ADR) | During the colonoscopy examination
  The percentage of colonoscopies when the adenoma was found
Advanced adenoma detection rate (AADR) | During the colonoscopy examination
  The percentage of colonoscopies when the advanced adenoma (>10mm) was found
Adenoma per colonoscopy score (APC) | During the colonoscopy examination
  The average number of adenomas detected in a single colonoscopy

SECONDARY OUTCOMES:
Laterally spreading tumor detection rate | During the colonoscopy examination
  The percentage of colonoscopies when the laterally spreading tumor lesion was found

CONTACTS AND LOCATIONS:
Overall Officials: Zofia Orzeszko, MD, Principal Investigator — Jagiellonian University; Miroslaw Szura, PhD, Prof., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spadaccini M, Iannone A, Maselli R, Badalamenti M, Desai M, Chandrasekar VT, Patel HK, Fugazza A, Pellegatta G, Galtieri PA, Lollo G, Carrara S, Anderloni A, Rex DK, Savevski V, Wallace MB, Bhandari P, Roesch T, Gralnek IM, Sharma P, Hassan C, Repici A. Computer-aided detection versus advanced imaging for detection of colorectal neoplasia: a systematic review and network meta-analysis. Lancet Gastroenterol Hepatol. 2021 Oct;6(10):793-802. doi: 10.1016/S2468-1253(21)00215-6. Epub 2021 Aug 5. PMID 34363763
- [Background] Barua I, Vinsard DG, Jodal HC, Loberg M, Kalager M, Holme O, Misawa M, Bretthauer M, Mori Y. Artificial intelligence for polyp detection during colonoscopy: a systematic review and meta-analysis. Endoscopy. 2021 Mar;53(3):277-284. doi: 10.1055/a-1201-7165. Epub 2020 Sep 29. PMID 32557490
- [Background] Repici A, Badalamenti M, Maselli R, Correale L, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Hassan C. Efficacy of Real-Time Computer-Aided Detection of Colorectal Neoplasia in a Randomized Trial. Gastroenterology. 2020 Aug;159(2):512-520.e7. doi: 10.1053/j.gastro.2020.04.062. Epub 2020 May 1. PMID 32371116
- [Background] Wang P, Liu P, Glissen Brown JR, Berzin TM, Zhou G, Lei S, Liu X, Li L, Xiao X. Lower Adenoma Miss Rate of Computer-Aided Detection-Assisted Colonoscopy vs Routine White-Light Colonoscopy in a Prospective Tandem Study. Gastroenterology. 2020 Oct;159(4):1252-1261.e5. doi: 10.1053/j.gastro.2020.06.023. Epub 2020 Jun 17. PMID 32562721
- [Background] Glissen Brown JR, Mansour NM, Wang P, Chuchuca MA, Minchenberg SB, Chandnani M, Liu L, Gross SA, Sengupta N, Berzin TM. Deep Learning Computer-aided Polyp Detection Reduces Adenoma Miss Rate: A United States Multi-center Randomized Tandem Colonoscopy Study (CADeT-CS Trial). Clin Gastroenterol Hepatol. 2022 Jul;20(7):1499-1507.e4. doi: 10.1016/j.cgh.2021.09.009. Epub 2021 Sep 14. PMID 34530161
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339